CLINICAL TRIAL: NCT06634953
Title: The Impact of Volleyball on Menstrual Symptoms in Adolescent Athletes
Brief Title: The Impact of Volleyball on Menstrual Symptoms
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Seda Uluşahin, PT PhD, Saglik Bilimleri Universitesi
Other Study IDs: 2023-1569
Record Dates: First submitted 2024-10-03; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Adolescent; Female; Menstruation
Keywords: volleyball; adolescent athlete; menstruation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescent female volleyball athletes: willingness to participate in the research, female gender, experience of menstruation cycles for at least 1 year, age between 10 and 19 years, volleyball sport license for at least 3 years, and practice of volleyball at least 4 days a week for at least 3 years
- Healthy adolescent females: willingness to participate in the research, female gender, experience of menstruation cycles for at least 1 year, age between 10 and 19 years,

SUMMARY:
The goal of this observational study is to examine menstrual characteristics and symptoms in adolescent volleyball athletes compared to non-athlete adolescents. The main question it aims to answer is:

How do menstrual symptoms and characteristics differ between adolescent volleyball athletes and non-athletes?

The study included 154 adolescents aged 10-19, divided into 77 volleyball athletes (average age 15.09) and 77 non-athletes (average age 14.79). Assessments covered menstruation age, regularity, dysmenorrhea characteristics, and menstrual symptoms using the Menstrual Symptom Questionnaire (MSQ).

DETAILED DESCRIPTION:
The goal of this observational study is to investigate menstrual characteristics and symptoms in adolescent volleyball athletes compared to non-athlete adolescents. The main question it aims to answer is:

How do menstrual symptoms and characteristics differ between adolescent volleyball athletes and their non-athlete peers?

The study included 154 adolescents aged 10-19 who had experienced menarche for at least one year. Participants were divided into two groups: 77 volleyball athletes (average age 15.09±1.33) and 77 non-athletes (average age 14.79±1.27). Assessments included menstruation age, regularity, use of menstruation delay pills, cycle characteristics (length, duration), and dysmenorrhea characteristics (onset, frequency, medication use, school/training absenteeism). The Menstrual Symptom Questionnaire (MSQ) evaluated menstrual pain, coping methods, and somatic complaints.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate in the research,
* female gender,
* experience of menstruation cycles for at least 1 year,
* age between 10 and 19 years,
* having a volleyball sport license for at least 3 years,
* practicing of volleyball at least 4 days a week for at least 3 years.

Exclusion Criteria:

* being pregnant
* experiencing acute genital infection
* gynecological or urological surgery
* having a diagnosis with an endocrine, systemic, or psychological disease.

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female
Study Population: 10-19 years old females
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Menstrual Pain | 3 months ( will cover 3 menstrual cyles)
  Menstruation related pain ( pain in the first 3 days of menstruation) intensity will be measured as a primary outcome using the the Visual Analog Scale (VAS). This outcome will measure the level of pain experienced by participants and the results will be reported as a continuous variable. The VAS consists of a 10 cm horizontal line with endpoints labeled "no pain" (0) and "worst pain imaginable" . Participants will mark the point on the line that best represents their pain intensity. The scores range from 0 (no pain) to 10 (worst pain), with higher scores indicating worse pain.
Menstrual symptoms (assessed using the Menstruation Symptom Questionnaire) | 3 months. The outcome will be evaluated before starting the study and after 12 weeks. It will be reported as a continuous variable to quantify changes in symptom severity over time.
  Menstrual symptoms will be assessed using the Menstruation Symptom Questionnaire (MSQ) designed to measure the severity and frequency of physical and emotional symptoms associated with menstruation (Negative Effects/Somatic Complaints, Menstrual Pain, and Coping Methods). The MSQ consists of 24 items, each rated on a 5-point Likert scale where 0 indicates no symptoms and 5 indicates the most severe symptoms.
  The total MSQ score ranges from 0 to 120, with higher scores reflecting worse menstrual symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Saglik Bilimleri Universitesi, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Participants datas will not be shared till publicaiton is confirmed